CLINICAL TRIAL: NCT02013570
Title: Efficacy of Peritonsillar Dexmedetomidine Infiltration for Postadenotonsillectomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Isin Gunes, Assistant Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/556
Record Dates: First submitted 2013-12-02; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-09

CONDITIONS: Pain Postoperative, Intraoperative Hemorrhage
Keywords: postoperative pain; dexmedetomidine; adenotonsillectomy
MeSH Terms: conditions — Pain, Postoperative; Blood Loss, Surgical | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dexmedetomidine (Active Comparator): Group S peritonsillar 2ml normal saline (1 ml per tonsil) via peritonsillar infiltration.
  Interventions: Drug: Dexmedetomidine
- Normal saline, postoperative pain (Placebo Comparator): Group S peritonsillar 2ml normal saline (1 ml per tonsil) via peritonsillar infiltration.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 2µg/kg dexmedetomidine in 2 ml normal saline (1 ml per tonsil),
  Other Names: Precedex

SUMMARY:
The purpose of the present study is the clinical assessment of the efficacy of preincisional peritonsillar infiltration of dexmedetomidine on postoperative pain relief in children undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Background:Tonsillectomy is a common and painful procedure in children, often performed on an outpatient basis. Tonsillectomy is often associated with intraoperative bleeding and postoperative severe pain. Different methods such as drugs (nonsteroidal antiinflammatory drugs , opioids, corticosteroids ), adjustment of surgical technique and peroperative local anaesthetic infiltration have been used to reduce pain. It is known that pain after adenotonsillectomy or analgesic usage may lead to unwanted effects. For example, nonsteroidal antiinflammatory drugs may interfere with bleeding and opioids may cause respiratory depression, sedation or nausea and vomiting. There are some reported complications seen infiltrations of local anaesthetics into tonsillar and adenoid beds. No studies have assessed the effects of peritonsillar dexmedetomidine infiltration. Dexmedetomidine is a centrally acting sympatholytic agent that has intrinsic effect of regional anesthesia with amid anesthetic.Because of its analgesic and sedating activity, dexmedetomidine has been used previously as an nasal premedication in patients undergoing tonsillectomy, but its use, as a peritonsillar infiltration has not been evaluated. Dexmedetomidine is a highly selective alfa-2 adrenoreceptor agonist recently introduced to anesthesia practice producing dose-depended sedation, anxiolysis, and analgesia (involving spinal and supraspinal sites), without respiratory depression. Also Alpha-2 adrenergic agonists have peripheral analgesic effects. Therefore, this study was designed to compare the effects of preincisional, dexmedetomidine 2µg/kg peritonsillar infiltration by peritonsillar normal saline grup on intraoperative bleeding and hemodynamics, postoperative recovery including pain, sedation, nausea and vomiting in pediatric patients undergoing adenotonsillectomy, and the recording of any adverse effects that might develop during the 24-h study period.

Methods: Seventy patient were randomized into two groups: group S peritonsillar 2ml normal saline (1 ml per tonsil), group D 2mikro gram/kg dexmedetomidine in 2 ml normal saline (1 ml per tonsil).

After institutional Ethics Committee approval and parents written consent, 70 children aged 3-9 years, American Society of Anesthesiologists 1-2 status, scheduled for adenotonsillectomy were enrolled in this randomized, prospective, triple-blind clinical study. Children with systemic disease, metabolic and endocrin disorders, growth developmental and motor-mental retardation, those who had a history of allergy to any of the study drugs, peritonsillar abscess, hypertension, psychiatric and epileptic disorders, chronic pain syndrome, and those who received analgesics within 24 h prior to surgery were excluded from study.

The children were unpremedicated. Anaesthesia was induced with sevoflurane 8% and nitrous oxide 70% in oxygen or intravenous induction with propofol (2,5-3 mg/kg). After induction rocuronium 0,6 mg/kg was administered for muscle relaxation and fentanyl 1 µg/kg before tracheal intubation. Anaesthesia was maintained with sevoflurane 2-3% and nitrous oxide 30% in oxygen. After intubation children were randomized into two groups:Group D 2µg/kg dexmedetomidine in 2 ml normal saline (1 ml per tonsil), Group S peritonsillar 2ml normal saline (1 ml per tonsil) via peritonsillar infiltration. For the infiltration, all injections were performed through the tonsillar capsule and anterior plica. After the infiltration, a minimum of 3 min was allowed for the onset of action of dexmedetomidine before adenotonsillectomy. Adenotonsillectomy was performed with snare technic by the same surgeon in all cases. Heart rate, arterial pressure and oxygen saturations (SpO2) were recorded at 10 min interval during operation.All patients received metoclopropamide 0,2 mg/kg i.v. before end of the surgery. After extubation the patients were taken to the postanesthesia care unit where an anesthetist and nurses who were unaware of the study drug observed the patients.

Modified Hannallah pain scale (observational pain scores-OPS), nausea, vomiting, bleeding, rescue analgesia, sedation and Aldrete scores were recorded on arrival in the postanesthesia care unit, at 15th, 30th, 60th, 90th and 120th min. Patient with OPS scores >4, for a patient request for pain medication, received 1mg/kg Tramadol drop as supplementary analgesia. The first analgesic requirement time recorded. Children vomiting twice or more in PACU received additional antiemetic drug (metoclopropamide 0,2 mg/kg i.v.). Agitation was measured with Pediatric anesthesia emergence delirium scale. Patients with an Aldrete score of 9 were transferred to the postoperative surgical ward.

Pain, nausea and vomiting, bleeding and sedation were assessed in the postoperative surgical ward at0,2,4,6h follow-up by the nurses who were trained fort he use of scores involved. Analgesic requirement were recorded. Pain was measured at rest and with swallowing. All patients were discharged at the and of the day and stayed home at night. Before the discharge, parents were given a prescription for acetaminophen (15 mg/kg oral dose) to be given when needs to analgesia. Postoperative pain during the first 24 h was assessed using a four-point scale: 0=no pain, 1=mild pain, 2=moderate pain, 3=severe pain by questioning their parents. Patients were interviewed on the day after surgery to asses the postoperative pain, vomiting, bleeding and rescue analgesia. Family satisfaction was assessed as follows: 1=poor; 2=good; 3=perfect.

ELIGIBILITY:
Inclusion Criteria:

children aged 3-9 years American Society of Anesthesiologists 1-2 status, scheduled for adenotonsillectomy

Exclusion Criteria:

Children with systemic disease, metabolic and endocrin disorders, growth developmental and motor-mental retardation, those who had a history of allergy to any of the study drugs, peritonsillar abscess, hypertension, psychiatric and epileptic disorders, chronic pain syndrome, and those who received analgesics within 24 h prior to surgery were excluded from study.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
post adenotonsillectomy pain | 24 hours
  Modified Hannallah pain scale, nausea, vomiting, bleeding, rescue analgesia, sedation and Aldrete scores were recorded on arrival in the postanesthesia care unit, at 15th, 30th, 60th, 90th and 120th min. Patient with pain scores >4, for a patient request for pain medication, received 1mg/kg Tramadol drop as supplementary analgesia. The first analgesic requirement time recorded. Agitation was measured with Pediatric anesthesia emergence delirium scale. Patients with an Aldrete score of 9 were transferred to the postoperative surgical ward.
  Pain, nausea and vomiting, bleeding and sedation were assessed in the postoperative surgical ward. Analgesic requirement were recorded. Pain was measured at rest and with swallowing. All patients were discharged at the end of the day and stayed home at night. Postoperative pain during the first 24 h was assessed using a four-point scale. Patients were interviewed on the day after surgery to ases.